CLINICAL TRIAL: NCT00060606
Title: Myelomeningocele Repair Randomized Trial
Brief Title: Management of Myelomeningocele Study (MOMS)
Acronym: MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Children's Hospital of Philadelphia (Other); Vanderbilt University Medical Center (Other); University of California, San Francisco (Other); University of Pittsburgh Medical Center (Other); University of Houston (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01HD041665 (NIH); U01HD068541 (NIH); U01HD41666 (Other Grant/Funding Number: NICHD); U01HD41667 (Other Grant/Funding Number: NICHD); U01HD41669 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2003-05-08; First posted 2003-05-09 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Meningomyelocele; Spinal Dysraphism
Keywords: Maternal fetal surgery; Fetal diagnosis; Myelomeningocele; Meningomyelocele; Open neural tube defect; ONTD; Spina bifida
MeSH Terms: conditions — Meningomyelocele; Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal Surgery Group (Experimental): Fetal surgery to close spina bifida defect prior to 26 weeks of gestation with delivery by C-Section at approximately 37 weeks of gestation.
  Interventions: Procedure: Prenatal Myelomeningocele Repair Surgery
- Postnatal Surgery Group (Active Comparator): Standard postnatal closure of the spina bifida defect when the baby is medically stable, usually within 48 hours of birth by C-section.
  Interventions: Procedure: Postnatal Myelomeningocele Repair Surgery

INTERVENTIONS:
Procedure: Prenatal Myelomeningocele Repair Surgery — Fetal surgery to repair spina bifida defect performed prior to 26 weeks of gestation with delivery by C-section at approximately 37 weeks of gestation.
  Arms: Prenatal Surgery Group
Procedure: Postnatal Myelomeningocele Repair Surgery — Standard postnatal surgical closure of the spina bifida defect
  Arms: Postnatal Surgery Group

SUMMARY:
Spina bifida (myelomeningocele) is a complex birth defect in which a portion of the spinal cord is not fully developed. The overlying bones and skin are incompletely formed and the underdeveloped area of the spinal cord is exposed on the surface of the back. Spina bifida defects are closed soon after birth to prevent further damage to the spinal cord and nerves. The Management of Myelomeningocele Study (MOMS) is a research study comparing two approaches to the treatment of babies with spina bifida: surgery before birth (prenatal surgery) and the standard closure, surgery after birth (postnatal surgery).

DETAILED DESCRIPTION:
Since 1997, more than 200 fetuses have had in utero closure of myelomeningocele by open maternal-fetal surgery. Preliminary clinical evidence suggests that this procedure reduces the incidence of shunt-dependent hydrocephalus and restores the cerebellum and brainstem to more normal configuration. However, clinical results of prenatal surgery for myelomeningocele are based on comparisons with historical controls and examine only efficacy, not safety. MOMS will determine if intrauterine repair of fetal myelomeningocele at 19 to 25 weeks of gestation improves outcomes as compared to standard postnatal repair. Outcomes assessed include death, the need for ventricular decompressive shunting by one year of life and neurologic function at 30 months of age.

One hundred eighty-three women, whose fetuses have spina bifida, were enrolled in the study and randomized to have either prenatal surgery or postnatal surgery. After a central screening process which included a medical record review, all women had an extensive baseline evaluation that included ultrasound, MRI, physical exam, social work evaluation, psychological screening, and education about spina bifida and prenatal surgery.

For women who were eligible following the central screening process, all screening, surgery and follow-up visits were performed at one of three MOMS Centers. The mother, if eligible, and her support person traveled (at the expense of the study) to the MOMS Center for screening and randomization.

Women assigned to have prenatal surgery were scheduled for surgery within 1 to 3 days after they were randomized. They stayed near the MOMS Center until they delivered. Women in the postnatal group traveled back to their assigned MOMS Center to deliver. Both groups delivered their babies by C-section around the 37th week of their pregnancies. Babies born to women in the postnatal surgery group had their spina bifida defects closed when they were medically stable, usually within 48 hours of birth.

Children and their parents returned to their assigned MOMS Center at 1 year and 2 ½ years of age for follow-up evaluation. Motor function, developmental progress, and bladder, kidney, and brain development were assessed.

The children were asked to return for an additional follow-up visit (MOMS2) between the ages of 6-10 years. This follow-up is to determine whether children who received the surgery before birth have better health and mental outcomes and live more independently and function more safely and appropriately in daily life than those who received the surgery after birth.

ELIGIBILITY:
Inclusion Criteria

* Pregnant women carrying a fetus diagnosed with myelomeningocele
* Myelomeningocele lesion that starts no higher than T1 and no lower than S1 with hindbrain herniation present
* Gestational age at randomization of 19 weeks 0 days to 25 weeks 6 days
* Normal karyotype
* Singleton pregnancy
* United States resident
* Able to travel to study site for study evaluation, procedures, and visits (if randomized to prenatal surgery, must stay near center until delivery)
* Support person to travel and stay with participant

Exclusion Criteria

* Maternal insulin-dependent pregestational diabetes
* Short or incompetent cervix or cervical cerclage
* Placenta previa
* Body mass index of 35 or more
* Previous spontaneous delivery prior to 37 weeks
* Maternal HIV, Hepatitis-B or Hepatitis-C status positive
* Uterine anomaly
* Maternal medical condition which is a contraindication to surgery or general anesthesia
* Other fetal anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2003-02; Primary Completion 2014-02 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Thom, PhD, Principal Investigator — George Washington University, Data and Study Coordinating Center
Locations (3):
- United States (3):
  - University of California at San Francisco, San Francisco, California
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses.

REFERENCES:
- [Result] Adzick NS, Thom EA, Spong CY, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Dabrowiak ME, Sutton LN, Gupta N, Tulipan NB, D'Alton ME, Farmer DL; MOMS Investigators. A randomized trial of prenatal versus postnatal repair of myelomeningocele. N Engl J Med. 2011 Mar 17;364(11):993-1004. doi: 10.1056/NEJMoa1014379. Epub 2011 Feb 9. PMID 21306277
- [Result] Tulipan N, Wellons JC 3rd, Thom EA, Gupta N, Sutton LN, Burrows PK, Farmer D, Walsh W, Johnson MP, Rand L, Tolivaisa S, D'alton ME, Adzick NS; MOMS Investigators. Prenatal surgery for myelomeningocele and the need for cerebrospinal fluid shunt placement. J Neurosurg Pediatr. 2015 Dec;16(6):613-20. doi: 10.3171/2015.7.PEDS15336. Epub 2015 Sep 15. PMID 26369371
- [Result] Brock JW 3rd, Carr MC, Adzick NS, Burrows PK, Thomas JC, Thom EA, Howell LJ, Farrell JA, Dabrowiak ME, Farmer DL, Cheng EY, Kropp BP, Caldamone AA, Bulas DI, Tolivaisa S, Baskin LS; MOMS Investigators. Bladder Function After Fetal Surgery for Myelomeningocele. Pediatrics. 2015 Oct;136(4):e906-13. doi: 10.1542/peds.2015-2114. PMID 26416930
- [Result] Johnson MP, Bennett KA, Rand L, Burrows PK, Thom EA, Howell LJ, Farrell JA, Dabrowiak ME, Brock JW 3rd, Farmer DL, Adzick NS; Management of Myelomeningocele Study Investigators. The Management of Myelomeningocele Study: obstetrical outcomes and risk factors for obstetrical complications following prenatal surgery. Am J Obstet Gynecol. 2016 Dec;215(6):778.e1-778.e9. doi: 10.1016/j.ajog.2016.07.052. Epub 2016 Aug 2. PMID 27496687
- [Result] Antiel RM, Adzick NS, Thom EA, Burrows PK, Farmer DL, Brock JW 3rd, Howell LJ, Farrell JA, Houtrow AJ; Management of Myelomeningocele Study Investigators. Impact on family and parental stress of prenatal vs postnatal repair of myelomeningocele. Am J Obstet Gynecol. 2016 Oct;215(4):522.e1-6. doi: 10.1016/j.ajog.2016.05.045. Epub 2016 Jun 2. PMID 27263997
- [Result] Farmer DL, Thom EA, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Gupta N, Adzick NS; Management of Myelomeningocele Study Investigators. The Management of Myelomeningocele Study: full cohort 30-month pediatric outcomes. Am J Obstet Gynecol. 2018 Feb;218(2):256.e1-256.e13. doi: 10.1016/j.ajog.2017.12.001. Epub 2017 Dec 12. PMID 29246577
- [Result] Brock JW 3rd, Thomas JC, Baskin LS, Zderic SA, Thom EA, Burrows PK, Lee H, Houtrow AJ, MacPherson C, Adzick NS; Eunice Kennedy Shriver NICHD MOMS Trial Group. Effect of Prenatal Repair of Myelomeningocele on Urological Outcomes at School Age. J Urol. 2019 Oct;202(4):812-818. doi: 10.1097/JU.0000000000000334. Epub 2019 Sep 6. PMID 31075056
- [Result] Houtrow AJ, Burrows PK, Thom EA. Comparing neurodevelopmental outcomes at 30 months by presence of hydrocephalus and shunt status among children enrolled in the MOMS trial. J Pediatr Rehabil Med. 2018;11(4):227-235. doi: 10.3233/PRM-170481. PMID 30507586
- [Result] Oliver ER, Heuer GG, Thom EA, Burrows PK, Didier RA, DeBari SE, Martin-Saavedra JS, Moldenhauer JS, Jatres J, Howell LJ, Adzick NS, Coleman BG. Myelomeningocele sac associated with worse lower-extremity neurological sequelae: evidence for prenatal neural stretch injury? Ultrasound Obstet Gynecol. 2020 Jun;55(6):740-746. doi: 10.1002/uog.21891. PMID 31613408
- [Derived] Houtrow AJ, MacPherson C, Jackson-Coty J, Rivera M, Flynn L, Burrows PK, Adzick NS, Fletcher J, Gupta N, Howell LJ, Brock JW 3rd, Lee H, Walker WO, Thom EA. Prenatal Repair and Physical Functioning Among Children With Myelomeningocele: A Secondary Analysis of a Randomized Clinical Trial. JAMA Pediatr. 2021 Apr 1;175(4):e205674. doi: 10.1001/jamapediatrics.2020.5674. Epub 2021 Apr 5. PMID 33555337
- [Derived] Swarup I, Talwar D, Howell LJ, Adzick NS, Horn BD. Orthopaedic outcomes of prenatal versus postnatal repair of myelomeningocele. J Pediatr Orthop B. 2022 Jan 1;31(1):87-92. doi: 10.1097/BPB.0000000000000827. PMID 33165214
- [Derived] Houtrow AJ, Thom EA, Fletcher JM, Burrows PK, Adzick NS, Thomas NH, Brock JW 3rd, Cooper T, Lee H, Bilaniuk L, Glenn OA, Pruthi S, MacPherson C, Farmer DL, Johnson MP, Howell LJ, Gupta N, Walker WO. Prenatal Repair of Myelomeningocele and School-age Functional Outcomes. Pediatrics. 2020 Feb;145(2):e20191544. doi: 10.1542/peds.2019-1544. PMID 31980545
- [Derived] Etchegaray A, Palma F, De Rosa R, Russo RD, Beruti E, Fregonese R, Allegrotti H, Musante G, Cibert A, Storz FC, Marchionatti S. [Fetal surgery for myelomeningocele: Obstetric evolution and short-term perinatal outcomes of a cohort of 21 cases]. Surg Neurol Int. 2018 Nov 26;9(Suppl 4):S73-S84. doi: 10.4103/sni.sni_236_18. eCollection 2018. Spanish. PMID 30595963

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prenatal Surgery Group | Postnatal Surgery Group
Started | 91 | 92
First Primary Outcome - Shunt at 12 Mont | 91 | 92
Completed (Second primary outcome - 30 months) | 91 | 91
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Postnatal Surgery Group: Postnatal Myelomeningocele Repair Surgery: Standard postnatal surgical closure of the spina bifida defect when the baby is medically stable, usually within 48 hours of birth by C-section.
- Total: Total of all reporting groups
Arm/Group | Prenatal Surgery Group | Postnatal Surgery Group | Total
Number analyzed (Participants) | 91 | 92 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (5.2) | 28.7 (4.8) | 28.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 92 | 183
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 85 | 86 | 171
  Black Non-Hispanic | 1 | 1 | 2
  Hispanic | 3 | 4 | 7
  Other | 2 | 1 | 3
Gestational Age at randomization [Mean (Standard Deviation); unit: weeks] | 23.7 (1.4) | 23.9 (1.3) | 23.8 (1.3)
Married [Count of Participants; unit: Participants] | 84 | 86 | 170
Schooling [Mean (Standard Deviation); unit: years] | 14.9 (1.7) | 14.9 (1.7) | 14.9 (1.7)
Body Mass Index at screening [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (3.7) | 26.3 (3.9) | 26.3 (3.8)
Severe hindbrain herniation [Count of Participants; unit: Participants] | 27 | 23 | 50
Clubfoot [Count of Participants; unit: Participants] | 24 | 19 | 43
Fetal sex female [Count of Participants; unit: Participants] | 42 | 57 | 99
Nullipara [Count of Participants; unit: Participants] — First pregnancy
  Participants | 37 | 37 | 74
Previous uterine surgeries [Count of Participants; unit: Participants] | 12 | 11 | 23
Cervical length (transvaginal) [Mean (Standard Deviation); unit: mm] | 39.5 (7.6) | 39.4 (5.9) | 39.5 (6.8)
Spina bifida lesion level L3 or lower [Count of Participants; unit: Participants] — screening ultrasound
  Participants | 62 | 76 | 138

OUTCOME MEASURES:

1. Primary Outcome: Infant Death or Need for Ventricular Shunt by 1 Year of Life
Time Frame: 12 months of age
Measure: Count of Participants; unit: Participants
Groups:
- Prenatal Surgery: Fetal surgery to close spina bifida defect prior to 26 weeks of gestation with delivery by C-Section at approximately 37 weeks of gestation.
  Prenatal Myelomeningocele Repair Surgery: Fetal surgery to repair spina bifida defect performed prior to 26 weeks of gestation with delivery by C-section at approximately 37 weeks of gestation.
- Postnatal Surgery: Standard postnatal closure of the spina bifida defect when the baby is medically stable, usually within 48 hours of birth by C-section.
  Postnatal Myelomeningocele Repair Surgery: Standard postnatal surgical closure of the spina bifida defect
Arm/Group | Prenatal Surgery | Postnatal Surgery
Number analyzed (Participants) | 91 | 92
Participants | 66 | 90

2. Primary Outcome: Bayley Scales of Infant Development MDI and the Difference Between the Functional and Anatomical Level of Lesion at 30 Months of Age
Description: Individual outcome score is the sum of the following:
  1. Rank for the Bayley score which was constructed from the Bayley Scales of Infant Development Mental Development Index standardized score for each child at 30 months. Deaths had the lowest score of 0, lower than the lowest standardized score of 49. Scores were then ranked from 1 to 182 (1 is worst,182 is best).
  2. Rank for the difference between the anatomic and functional lesion levels of the spine was generated by a plain x-ray obtained at the 12-month visit for the anatomic level and the physical examination at 30 months for the functional level. The difference between the two was calculated where a positive difference means that the child is functioning better than expected by the level of his/her lesion. Deaths received the lowest score of -25, lower than all other possible differences. The differences were then ranked from 1 to 182 (1 is worst, 182 is best).
  For the overall score, 2 is the worst and 364 is the best.
Time Frame: 30 months of age
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prenatal Surgery | Postnatal Surgery
Number analyzed (Participants) | 91 | 91
units on a scale | 199.4 (80.5) | 166.6 (76.7)

3. Secondary Outcome: Number of Participants Walking Independently at Examination
Time Frame: 30 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Surgery | Postnatal Surgery
Number analyzed (Participants) | 87 | 88
Participants | 39 | 21

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of randomization through 30 months of life.
Arm/Group | Prenatal Surgery Group | Postnatal Surgery Group
All-Cause Mortality (participants affected / at risk) | 4/91 | 3/92
Serious Adverse Events (participants affected / at risk) | 4/91 | 3/92
Other Adverse Events (participants affected / at risk) | 0/91 | 0/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prenatal Surgery Group (N=91) | Postnatal Surgery Group (N=92)
Fetal or infant death (General disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less